CLINICAL TRIAL: NCT00000649
Title: An Open-Label, Staggered Rising Dose Cohort Study Assessing the Pharmacokinetics, Safety, and Tolerance of BI-RG-587 in Combination With Zidovudine in Patients With HIV Infection (CD4+ Cell Count < 400/mm3)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Organization: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG 168; 00834
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 1993-06

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Nevirapine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nevirapine; Zidovudine

INTERVENTIONS:
Drug: Nevirapine
Drug: Zidovudine

SUMMARY:
To assess the safety and tolerance of multiple oral doses of nevirapine in combination with zidovudine (AZT); to get information on the pharmacokinetics (blood levels) and dose proportionality of nevirapine/AZT with multiple dosing; to characterize the pattern of virological activity in vivo (in humans) of nevirapine in combination with AZT; to determine whether development of resistance to either drug is slowed by the use of the combination.

Drugs now used in treatment for patients with AIDS show some toxicity which limits their usefulness. In addition, with long-term treatment with AZT, there is evidence of virus resistance to the drug. Compounds that are more effective and less toxic than those in present use would be beneficial, especially if they are active against AZT-resistant viruses. Nevirapine has shown in vitro (test tube studies) activity in inhibiting HIV replication (reproduction). In vitro studies have shown that nevirapine and AZT work together to inhibit HIV replication.

DETAILED DESCRIPTION:
Drugs now used in treatment for patients with AIDS show some toxicity which limits their usefulness. In addition, with long-term treatment with AZT, there is evidence of virus resistance to the drug. Compounds that are more effective and less toxic than those in present use would be beneficial, especially if they are active against AZT-resistant viruses. Nevirapine has shown in vitro (test tube studies) activity in inhibiting HIV replication (reproduction). In vitro studies have shown that nevirapine and AZT work together to inhibit HIV replication.

Groups of 10 patients are studied at each of three dose levels. Five patients at each dose level have less than 3 months of prior AZT treatment; five patients at each dose level have at least 12 months of previous AZT treatment and tolerated an AZT regimen of 600 mg/day (200 mg every 8 hours). At least 24 patient-weeks of treatment with the combination treatment must be completed without requiring dose interruption before the next dosage level can be started. All 30 patients must be enrolled at a lower dosage level before a higher dosage level is started. Patients begin treatment with AZT. 14 days later, patients begin treatment with nevirapine in addition to the AZT. After 24 weeks, patients have the option to continue long-term treatment with either nevirapine or standard treatment.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication: Included:

Pneumocystis carinii pneumonia prophylaxis (other than sulfamethoxazole alone or in combination with other medications).

* Antifungal prophylaxis with oral fluconazole or ketoconazole.
* Antiviral prophylaxis with a maximum of 1 g/day oral acyclovir.

Patients must have the following:

* HIV infection.
* Ability to voluntarily provide written informed consent prior to treatment.
* Willing and able to follow protocol requirements.
* Patients with nonvisceral Kaposi's sarcoma or with visceral Kaposi's sarcoma not requiring chemotherapy and/or irradiation may be included.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Radiographic evidence of chronic pulmonary disease.
* Cytomegalovirus disease.
* Toxoplasmosis encephalitis requiring suppressive therapy.
* Mycobacteriosis requiring maintenance chemotherapy.
* Visceral Kaposi's sarcoma requiring chemotherapy and/or irradiation.

Concurrent Medication:

Excluded:

* Glucocorticoids and steroid hormones (including oral contraceptives).
* Dicumarol, warfarin, and other anticoagulant medications.
* Nitroglycerin.
* Digitoxin.
* Valproic acid.
* Tolbutamide.
* Doxycycline.
* Chloramphenicol.
* Isoniazid.
* Antiepileptics (Phenobarbital and other barbiturates).
* Sulfonamides.

Excluded for up to 4 hours before and 4 hours after administration of drug 2:

* Antacids.
* Cimetidine.
* Carafate.
* Cholestyramine resin.
* Alcohol and alcohol-containing substances.
* Benzodiazepines (diazepam, triazolam).

Patients with the following are excluded:

* History of clinically important disease (defined as a disease that, in the opinion of the investigator, may either put the patient at risk because of participation in the study or a disease that may influence the results of the study or the patient's ability to participate in the study) other than HIV infection.
* Malignancy other than Kaposi's sarcoma or limited cutaneous basal cell carcinoma.

Prior Medication:

Excluded within 4 weeks prior to administration of study drug 2:

* Antiretroviral (other than zidovudine (AZT)), immunosuppressive, or cytotoxic drugs.
* Glucocorticoids and steroid hormones (including oral contraceptives).
* Dicumarol, warfarin, and other anticoagulant medications.
* Nitroglycerin.
* Digitoxin.
* Valproic acid.
* Tolbutamide.
* Doxycycline.
* Chloramphenicol Isoniazid.
* Antiepileptics (Phenobarbital and other barbiturates).
* Sulfonamides.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Cheeseman, Study Chair
Locations (3):
- United States (3):
  - Cooper Green Hosp, Birmingham, Alabama
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Univ of Massachusetts, Worcester, Massachusetts

REFERENCES:
- [Background] Cheeseman SH. Nevirapine (NVP) alone and in combination with zidovudine (ZDV): safety and activity. The ACTG 164/168 Study Team. Int Conf AIDS. 1992 Jul 19-24;8(1):Mo15 (abstract no MoB 0053)
- [Background] Cheeseman SH, Havlir D, McLaughlin MM, Greenough TC, Sullivan JL, Hall D, Hattox SE, Spector SA, Stein DS, Myers M, et al. Phase I/II evaluation of nevirapine alone and in combination with zidovudine for infection with human immunodeficiency virus. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Feb 1;8(2):141-51. PMID 7530585
- [Background] Murphy RL, Montaner J. Nevirapine: A review of its development, pharmacological profile and potential for clinical use. Exp Opin Invest Drugs. 1996;5(9): 1183-1199
- [Background] Havlir D. Antiviral activity of nevirapine at 400 mg in p24 antigen positive adults. ACTG 164 and 168 Study Teams. Int Conf AIDS. 1993 Jun 6-11;9(1):69 (abstract no WS-B26-1)
- [Background] Greenough TC. Quantitative virology: the experience during the nevirapine phase I/II trials. ACTG 164/168 Study Team. Int Conf AIDS. 1992 Jul 19-24;8(2):B192 (abstract no PoB 3610)
- [Background] Cheeseman SH, Murphy RL, Saag MS, Havlir D. Safety of high dose nevirapine (NVP) after 200 mg/d lead-in. ACTG 164/168 Study Team. Int Conf AIDS. 1993 Jun 6-11;9(1):487 (abstract no PO-B26-2109)
- [Background] Hattox S. Pharmacokinetics of nevirapine alone and in combination with zidovudine. The ACTG 164/168 Study Team. Int Conf AIDS. 1992 Jul 19-24;8(2):B185 (abstract no PoB 3591)
- [Background] Richman DD. Loss of nevirapine activity associated with the emergence of resistance in clinical trials. The ACTG 164/168 Study Team. Int Conf AIDS. 1992 Jul 19-24;8(2):B183 (abstract no PoB 3576)